CLINICAL TRIAL: NCT01491321
Title: Clinical Trial to Evaluate the Efficacy of Bee Venom Acupuncture on Chronic Low Back Pain
Brief Title: Bee Venom Acupuncture for the Treatment of Chronic Low Back Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, JLee, Clinical Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2011-006
Record Dates: First submitted 2011-12-07; First posted 2011-12-14 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; bee venom acupuncture
MeSH Terms: interventions — loxoprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Bee Venom Acupuncture & Loxoprofen (Experimental)
  Interventions: Procedure: Bee Venom Acupuncture Therapy; Drug: Loxoprofen
- Sham Bee Venom Acupuncture & Loxoprofen (Placebo Comparator)
  Interventions: Drug: Loxoprofen; Procedure: Placebo

INTERVENTIONS:
Procedure: Bee Venom Acupuncture Therapy — Bee Venom 1:20,000 under BVA Increment Protocol
  Increment Protocol as
  * 1st week : SC 0.2cc/day, 2days/week
  * 2nd week : SC 0.4cc/day, 2days/week
  * 3rd week : SC 0.8cc/day, 2days/week
  Other Names: pharmacopuncture
  Arms: Bee Venom Acupuncture & Loxoprofen
Drug: Loxoprofen — 60 mg/Tab, pers os 1Tab tid, for 3 weeks
  Other Names: Loxonin
Procedure: Placebo — Normal Saline (0.9% NaCl) under NS Increment Protocol
  Increment Protocol as
  * 1st week : SC 0.2cc/day, 2days/week
  * 2nd week : SC 0.4cc/day, 2days/week
  * 3rd week : SC 0.8cc/day, 2days/week
  Arms: Sham Bee Venom Acupuncture & Loxoprofen

SUMMARY:
The purpose of this study is to evaluate the efficacy of bee venom acupuncture on pain intensity, functional status and quality of life of patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* nonspecific, chronic low back pain over 3 months
* Must have LBP of more than VAS 4

Exclusion Criteria:

* cancer, vertebral fracture, spinal infection, inflammatory spondylitis
* spinal operation
* radicular pain
* other musculoskeletal pain
* physicological or mental disorders
* allergic history to BV therapy or insect bite

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for bothersomeness | Changes from baseline in VAS at 1 month

SECONDARY OUTCOMES:
Visual Analogue Scale for pain intensity | Changes from baseline in VAS at 1 month
Disability scores on Oswestry Disability Index | Changes from baseline in ODI at 1 month
Quality of Life scores on EQ-5D | Changes from baseline in EQ-5D at 1 month
Depression scores on Beck Depression Inventory | Changes from baseline in BDI at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hwan Lee, Principal Investigator — Spine Center, Kyung Hee University Hospital at Gangdong; Byung-Kwan Seo, Study Director — Spine Center, Kyung Hee University Hospital at Gangdong; Dae-Jin Cho, Study Director — Spine Center, Kyung Hee University Hospital at Gangdong
Locations (1):
- Spine Center, Kyung Hee University Hospital at Gangdong, Seoul, South Korea

REFERENCES:
- [Derived] Seo BK, Lee JH, Sung WS, Song EM, Jo DJ. Bee venom acupuncture for the treatment of chronic low back pain: study protocol for a randomized, double-blinded, sham-controlled trial. Trials. 2013 Jan 14;14:16. doi: 10.1186/1745-6215-14-16. PMID 23317340